CLINICAL TRIAL: NCT00240604
Title: Treatment With Rosiglitazone for the Prevention of Glucose Intolerance in Patients Treated With Corticosteroids
Brief Title: Prevention of Corticosteroid-induced Glucose Intolerance
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Motti Muszkat, MD, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 7-29.10.04-HMO-CTIL
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Glucose Intolerance
Keywords: corticosteroid treatment; inflammatory diseases
MeSH Terms: conditions — Glucose Intolerance | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Rosiglitazone — 4 mg rosiglitazone per day

SUMMARY:
Glucose intolerance is frequent and serious complication of corticosteroid therapy. the aim of the study is to examine the hypothesis that co treatment with rosiglitazone can prevent glucose intolerance in patients treated with corticosteroids.

DETAILED DESCRIPTION:
Glucose intolerance is frequent and serious complication of corticosteroid therapy. the aim of the study is to examine the hypothesis that co treatment with rosiglitazone can prevent glucose intolerance in patients treated with corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* corticosteroid treatment

Exclusion Criteria:

* congestive heart failure pedal edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-04; Primary Completion 2013-12 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
plasma glucose concentration | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Arie BenYehuda, MD, Study Director — Hadassah University Hospital
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel